CLINICAL TRIAL: NCT04795999
Title: Opportunities Beyond the Narrative: An Intervention for Justice-Involved Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WestEd (Other)
Collaborators: Urban Strategies (Unknown); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jonathan Nakamoto, Senior Research Associate, WestEd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-03-4
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Study Will Examine the Impact of Project With

STUDY DESIGN:
Intervention Model Description: The treatment condition involves participation in a teen pregnancy prevention program, Project With. The comparison condition for the study is treatment as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project With program (Experimental): Project With is a 12-lesson literary-based curriculum, delivered by Youth Advocates to youth in juvenile justice facilities and group homes in Southern California either in person or virtually, under COVID-19 contingencies. Program schedule is determined by the facility. The goals of Project With are to promote optimal health and reduce teen pregnancy and sexually transmitted infections (STIs).
  Interventions: Behavioral: Project With
- Treatment as usual (No Intervention): The counterfactual condition for the study is a business-as-usual condition.

INTERVENTIONS:
Behavioral: Project With — There are 12 lessons in Project With, typically delivered in six weekly sessions, with each session having two one-hour long lessons and a meal with facilitators in between the two lessons. Each lesson includes a discussion of selected literary works, including poetry, short stories, and excerpts from films and other videos. The curriculum is intended to be delivered to groups of 8-12 youth. In ideal program delivery, participants also share a meal with each other and with the Youth Advocate. Shared mealtimes create group cohesion and allow Youth Advocates to connect with participants on a personal level, building trust. At the end of the Project With curriculum, youth will partake in an offsite day excursion to Camp Eaton, a wooded camp outside of Los Angeles. At Camp Eaton, Youth Advocates will lead a Project With session, lunch, bonding activities and games, and an opportunity to engage in an outdoor activity.
  Arms: Project With program

SUMMARY:
WestEd and its partners Urban Strategies, the Los Angeles County Probation Department, Boys Republic, California Family Life Center, and Eggleston Youth Centers Inc. are conducting a quasi-experimental design to evaluate an innovative teen pregnancy prevention program, Project With, for incarcerated and other justice-involved youth in Southern California. Project With is a 12-lesson literary-based curriculum that utilizes group discussions of literary works and films to address personal relationships and sexual health topics. This study involves youth (age 15-19) at high risk for involvement in risky sexual behaviors, including teen pregnancy. The intervention shows potential to promote optimal health and reduce teen pregnancy and sexually transmitted infections (STIs) among incarcerated and other justice-involved youth, based on a previous formative evaluation of the intervention in 2018-2020. The purpose of this study is to test the curriculum on a population of incarcerated and other justice-involved youth.

DETAILED DESCRIPTION:
Urban Strategies was funded by a Teen Pregnancy Prevention (TPP) grant from the Office of Population Affairs (OPA) within the Department of Health and Human Services (DHHS) to conduct a rigorous evaluation of a TPP program, Project With, to determine the impact of this innovative literary-based curriculum for incarcerated and other justice-involved youth. Project With is a 12-lesson literary-based curriculum, typically delivered in six weekly sessions, with each session having two one-hour long lessons and a meal with facilitators in between the two lessons. Each lesson includes a discussion of selected literary works, including poetry, short stories, and excerpts from films and other videos. The intervention shows potential to promote optimal health and reduce teen pregnancy and sexually transmitted infections (STIs) among incarcerated and other justice-involved youth. This intervention builds upon a former TPP grant. A formative evaluation of the intervention with OPA funding was carried out from 2018-2020. The formative evaluation showed that the curriculum, which explores healthy and unhealthy relationships as they appear within literary works and is facilitated by a caring mentor using a culturally attuned approach, deeply engages incarcerated youth.

This study involves youth aged 15-19 who are incarcerated/justice-involved and who are at high risk for involvement in risky sexual behaviors, including teen pregnancy. The findings from this study are intended to contribute to research on teen pregnancy, sexual health, and healthy relationships. The population of justice-involved/incarcerated youth face historical, structural, and environmental factors that bring about distressing sexual health disparities. Nationwide, 20% of incarcerated youth already have a child or are either pregnant or expecting a child they fathered (Sedlak & Bruce, 2016). Rates of teen fatherhood for incarcerated youth are seven times higher than their peers, and rates of teen motherhood for incarcerated girls are one-third higher than national averages. Along with disparities related to teen pregnancy, incarcerated youth have high rates of trauma, thus any intervention for these youth must be trauma-informed. A 2010 Office of Juvenile Justice and Delinquency Prevention (OJJDP) report on the needs of incarcerated youth found 70% of all youth had experienced at least one childhood trauma, and 30% had experienced physical abuse, sexual abuse, or both. This study was designed to contribute to our understanding of what works with this population and to strengthen our knowledge base around developing and implementing a sexual health and personal relationships program.

The study will roll out in waves. During each wave a cohort of 8-12 youth from each facility will participate in Project With. After Urban Strategies implements Project With in a given facility, they will wait a period of time (e.g., one week to several months) and will then implement the program with a new cohort of youth. Using this design, each facility will participate in the study multiple times.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-19
* Residing in one of the Los Angeles County Probation Department camps or group homes within a partnered network
* Have the cognitive ability to complete the baseline and follow-up surveys in English or Spanish
* Need to be at the facilities for at least 8 weeks to complete the program

Exclusion Criteria:

* Outside of age criteria
* Not residing in one of the Los Angeles County Probation Department camps or group homes within a partnered network
* Does not have the cognitive ability to complete the baseline and follow-up surveys in English or Spanish
* Not remaining at the facilities for 8 weeks or more
* Youth who participated in a previous evaluation wave as part of the treatment or comparison group cannot participate in the evaluation a second time (i.e., during a second wave)

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 415 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Risky sexual behaviors | Six months after the baseline
  The outcome will be assessed with three items that assess whether youth had sexual intercourse with multiple partners, sexual intercourse without a condom, and sexual intercourse without using any method of birth control in the past three months (Rotz et al., 2016).

SECONDARY OUTCOMES:
Ability to resist temptations and provocations | Two and six months after the baseline
  The outcome will be measured with six items from Svensson et al.'s (2010) seven-item scale. The items (e.g., "I get angry very fast.") have shown good reliability with youth aged 12 to 17 (α = .78; Svensson et al., 2010) and will be rated on a scale from 1 (not like me at all) to 5 (very much like me).
Planfulness | Two and six months after the baseline
  The outcome will be measured with a slightly modified version of Wills et al.'s (2007) six-item scale. The items (e.g., "I like to plan things ahead of time.") showed acceptable reliability (α = .73; Wills et al., 2007) with a sample of ninth graders and the items will be rated on a scale from 1 (not like me at all) to 5 (very much like me).
Acceptance of intimate partner violence | Two and six months after the baseline
  The outcome will be measured with the five-item general violence subscale from the Acceptance of Couple Violence Scale (McRae et al., 2018). The items (e.g., "There are times when violence between dating partners is okay.") in the subscale showed excellent reliability with a sample of young adults (α = .93; McRae et al., 2018) and will be rated on a scale from 1 (strongly disagree) to 5 (strongly agree).
Self-efficacy to avoid risky sexual behavior | Two and six months after the baseline
  The outcome will be measured with a modified version of the Galavotti et al. (1995) Condom Use Self-Efficacy Scale that measures self-efficacy for condom use. The scale includes five items that ask the respondent to indicate how sure they are that they would be able to use a condom in a range of situations (e.g., "If you have been using alcohol or other drugs...?"). The items will be rated on a 1 (not at all sure) to 5 (very sure) scale. Galavotti et al.'s (1995) Condom Use Self-Efficacy Scale showed high reliability with a sample of young adults (α = .88).
Intentions to engage in risky sexual behavior | Two and six months after the baseline
  The outcome will be measured with three items that were TPP performance measures. The items will assess whether the youth intend in the next year to 1) have sexual intercourse, 2) use a condom if they have sex, and 3) use any effective method of birth control if they have sex. The three items will be rated on a 1 (no, definitely not) to 4 (yes, definitely).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Nakamoto, PhD, Principal Investigator — WestEd
Locations (1):
- Urban Strategies, Alhambra, California, United States

IPD SHARING:
Plan to Share IPD: No